CLINICAL TRIAL: NCT05823610
Title: Intrapartum Ultrasonography in Evaluation of the Progress of Labor
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Other Study IDs: IPUS
Record Dates: First submitted 2023-04-09; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Progress pf Labor
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: The ultrasound parameters to be collected included the angle of progression, head-perineum distance and head-symphysis distance at rest and while pushing during contraction and the data between measurements taken at rest and while pushing. Also anatomical scanning for the episiotomy, perineal tears and obstetric anal sphincter injuries (OASI), also trauma to the levator ani muscle. All demographic, clinical and ultrasound variables were compared between women who had a spontaneous vaginal delivery (SVD) and those who eventually had an operative delivery (OD), vacuum -assisted or cesarean section (CS).
  Interventions: Diagnostic Test: ultrasound

INTERVENTIONS:
Diagnostic Test: ultrasound — The ultrasound parameters to be collected included the angle of progression, head-perineum distance and head-symphysis distance at rest and while pushing during contraction and the data between measurements taken at rest and while pushing. Also anatomical scanning for the episiotomy, perineal tears and obstetric anal sphincter injuries (OASI), also trauma to the levator ani muscle. All demographic, clinical and ultrasound variables were compared between women who had a spontaneous vaginal delivery (SVD) and those who eventually had an operative delivery (OD), vacuum -assisted or cesarean section (CS).

SUMMARY:
The optimal management of the second stage of labor is a subject of an ongoing debate. It is well established that prolonged second stage of labor is associated with increased maternal and neonatal morbidity.

Diagnosing the onset of labour is one of the most critical and complex judgments made by care providers in the delivery room. Measurement of cervical dilatation is considered the most crucial parameter for labour progress during childbirth and the main reason for doing digital vaginal examination (DVE) in women with signs of labour onset.

DVE was the most common method for measuring cervical dilatation in the past and has been the gold standard for assessing labour progress. However, it can be subjective, inaccurate, and uncomfortable for women. Also, only 50% of assessments are accurate, and there is an increased risk of infection with frequent DVE. Therefore, vaginal examination cannot be a correct scale for measuring cervical dilatation, mainly when done by different examiners. Because of the poor reliability and pain associated with DVE, the use of intrapartum ultrasound to measure cervical dilation has been suggested as an alternative method. Abdominal, vaginal, trans-labial, and trans-perineal 2D and 3D ultrasounds have been used to measure cervical dilatation during labour.

ELIGIBILITY:
Inclusion Criteria:

* Primigravida patients
* At the onset of active phase
* Cephalic vertex presentation
* Estimated Fetal Weight 3Kg - 4Kg
* Gestational Age ≥37 weeks

Exclusion Criteria:

* Multiple Pregnancy
* Patients refused to participate in our study
* Induced labor
* Any Obstetrical Complication or Disease
* Malpresentation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: women presented in labor
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
compare the intrapartum sonographic parameters between women who had spontaneous vaginal delivery (SVD) vs those who required CS | one hour
  Ultrasound evaluation of the parameters of progress of labour